CLINICAL TRIAL: NCT05414058
Title: Adjunctive Methylphenidate Extended Release in Patients With Schizophrenia: a Single-centre Fixed Dose Cross-over Open-label Trial to Improve Functional and Cognitive Outcomes
Brief Title: Adjunctive Methylphenidate ER in Patients With Schizophrenia to Improve Functional and Cognitive Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021025
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia Schizoaffective
Keywords: schizophrenia; methylphenidate; functional outcomes
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: An open-label fixed dose controlled cross-over trial is planned. Participants will be randomized into one of two arms: 1) participants will receive four weeks of add-on methylphenidate ER 36 mg, or 2) participants will receive 4 weeks of treatment as usual (no-treatment control group). At 4 weeks, participants will switch arms for another 4 weeks.
Masking Description: An open-label fixed dose controlled cross-over trial is planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apo-Methylphenidate ER arm (Experimental): Apo-Methylphenidate ER, 36 mg, oral, once a day, every morning, 4 weeks duration. Methylphenidate ER will be started at 18 mg to test tolerability and will be titrated at day 7 to a dose of 36 mg.
  Interventions: Drug: Apo-Methylphenidate ER
- Treatment as usual arm (No Intervention): Participants in the treatment as usual arm will continue with their current treatment as decided by their treatment team.

INTERVENTIONS:
Drug: Apo-Methylphenidate ER — For inpatients, the study medication will be administered by unit nurses, alongside their other medications. For outpatients, the study medication will be dispensed to the participant by the research assistant during their weekly visit. Patients will continue their regular medications as per standard of care.
  Arms: Apo-Methylphenidate ER arm

SUMMARY:
Two of the major features of schizophrenia spectrum illness, negative and cognitive symptoms, have been associated with poor functional outcome and burden of illness. Given the proposed role of dopaminergic hypoactivity, augmentation with psychostimulants has been postulated as one of the potential treatment options for negative and/or cognitive symptoms of schizophrenia. The major drawback for use of these agents is a potential risk of relapse or worsening of psychosis through direct or indirect dopamine agonism activity and a great deal of caution has been called for use of stimulants in individuals with psychosis. However, preliminary results of earlier studies indicated improvement of negative and cognitive symptoms with off-label use of adjunctive psychostimulants. The present study aims to assess off-label use of adjunct psychostimulants in patients with schizophrenia in a tertiary mental health centre, focusing on efficacy and safety.

DETAILED DESCRIPTION:
This project focuses on assessing efficacy of off-label use of adjunctive methylphenidate ER 36 mg among 24 stable patients with schizophrenia spectrum illness. This is a single centre study at the Royal Ottawa Mental Health Centre, Ottawa, Canada. An open-label fixed dose controlled cross-over trial is planned. Individuals (inpatients and outpatients) with schizophrenia who are stable on antipsychotic medications will be invited to participate in the study. Participants will be randomized into receiving four weeks of methylphenidate extended release (ER) 36 mg or treatment as usual and will switch group assignments for another 4 weeks. The duration of the study is 12 weeks for each participant, including 8 weeks of treatment (4 weeks treatment as usual and 4 weeks treatment as usual + adjunctive methylphenidate ER) and a follow-up visit at 12 weeks (study end point). A number of standardized scales will be used to measure functional capacity, cognition and symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Adult between the ages of 18-55; we chose an upper age limit of 55 years to exclude patients with potential age-related cognitive impairments which usually occur about a decade earlier in patients with schizophrenia
* Inpatient or outpatient with schizophrenia spectrum illness, on any antipsychotic medication
* Clinically stable for the past 4 weeks
* Able to communicate in English

Exclusion Criteria:

* Have known sensitivity to methylphenidate ER, as documented in the electronic medical record OR, as reported by the patient AND verified by pharmacy
* Have had treatment with ECT in the past 6 months
* Have a history of traumatic brain injury
* Have a contraindication to psychostimulants including:

  1. Uncontrolled hypertension
  2. Significant cardiovascular abnormality including history of cardiac interventions, history of myocardial infarction, unstable arrhythmia, congenital heart disease
  3. Known family history of premature cardiac death (for males <45, females <55)
  4. Known history of glaucoma
* Are currently pregnant or planning to become pregnant- a rapid urine pregnancy test will be done for female participants, and a refusal to take the test or a positive test will exclude the participant
* Have a diagnosis of substance induced psychosis
* Have any of the following diagnoses: neurodevelopmental delay, intellectual disability or neurocognitive disorder (dementia)
* Have a diagnosis of another currently significant and unstable psychiatric condition (i.e. depressive episode, active substance use disorder, etc.)
* Have a history of previous safety concerns directly driven by positive symptoms (e.g history of suicide attempt as directed by auditory hallucinations)
* Have current active suicidality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Defined as change in functioning | VRFCAT will be implemented at baseline, week 4, 8 and at follow-up at week 12.
  Change in functioning will be measured using the Virtual Reality Functional Capacity Assessment (VRFCAT) tool. The VRCAT is an interactive computerized measure of functional capacity. It presents the user with real life scenarios such as shopping, taking a bus, completing a recipe, etc, and assesses key instrumental activities of daily living in a realistic and interactive virtual environment.

SECONDARY OUTCOMES:
Defined as change in cognitive functioning (domains include verbal memory, working memory, motor speed, attention and processing speed, verbal fluency and executive functioning) | BACS will be implemented at baseline, week 4, 8 and at follow-up at week 12.
  Change in cognitive functioning will be measured using the Brief Assessment of Cognition in Schizophrenia (BACS). The BACS is a tool to assess aspects of cognition found to be the most impaired and correlated with outcome in patients with schizophrenia. It consists of six domains: verbal memory, working memory, motor speed, attention and processing speed, verbal fluency and executive functioning.

OTHER OUTCOMES:
Defined as symptom severity (items include delusions, conceptual disorganization, hallucinations, blunted affect, social withdrawal, lack of spontaneity/flow of conversation) | The PANSS-6 will be completed at all time points (baseline, weeks 1-8, and at follow-up at week 12.
  Symptom severity will be measured using the Positive and Negative Syndrome Scale 6-item (PANSS-6). The PANSS-6 is a 6-item version of the PANSS scale, and includes P1 = delusions, P2 = conceptual disorganization, P3 = hallucinations, N1 = blunted affect, N4 = social withdrawal, N6 = lack of spontaneity/flow of conversation. Items are rated on a 7-point scale from 1(absent) to 7(extreme), with a total range of 6-42, with higher scores indicative of more severe symptoms. The PANSS-6 has been shown to adequately measure severity, remission, and antipsychotic efficacy related to core positive and negative symptoms in clinical trials and its validity and sensitivity have been demonstrated in treatment resistant schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Naista Zhand, M.D., Principal Investigator — Royal Ottawa Mental Health Centre
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No